CLINICAL TRIAL: NCT05735054
Title: A Novel Technique for Endoscopic Transaxillary Thyroidectomy: a Preliminary Report and Comparison With the Open Procedure
Brief Title: A Novel Technique for Endoscopic Transaxillary Thyroidectomy Comparison
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 202303
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Thyroid Diseases
Keywords: endoscopy; thyroidectomy; transaxillary; open
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endoscopic group: the patients who underwent endoscopic transaxillary thyroidectomy
  Interventions: Procedure: endoscopic thyroidectomy
- open group: the patients who underwent open thyroidectomy
  Interventions: Procedure: endoscopic thyroidectomy

INTERVENTIONS:
Procedure: endoscopic thyroidectomy — the patients who underwent endoscopic transaxillary thyroidectomy

SUMMARY:
The clinical data from all except the first 20 cases who underwent our novel transaxillary thyroidectomy were collected retrospectively, while the data from patients who underwent conventional open thyroid lobectomy by same surgeon during the same period were used as a control.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with benign or malignant thyroid disease require lobe thyroidectomy;
2. The patient had cosmetic requirements and agreed with transaxillary thyroidectomy;
3. Benign lesions with the largest diameter ≤5 cm;
4. Differentiated thyroid cancer(DTC) meets the following conditions at the same time: ①The maximum diameter of the primary lesion is <2.5 cm; ②There is no extraglandular invasion or only minimal external invasion of the anterior thyroid capsule or minor invasion of the sternum thyroid muscle;

Exclusion Criteria:

1. the patients had poor compliance and could not be reexamined regularly;
2. There was a history of neck or thyroid surgery;
3. The patients require total thyroidectomy or lateral neck dissection.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the patient who required thyroidectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
operation time (OT) | during the operation
  The time will be reported as minutes.
bleeding | during the operation
  intraoperatively bleeding volume. The intraoperative blood lose volume will be reported as ml.
complications | 6 moths after oepration
  any complications after operation

SECONDARY OUTCOMES:
hospital stay | 1 week
  How many days will the patients stay in the hospital. The index will be reported as days.
drainage days. | 1 week
  This index will record how many days does the drainage tube keep in the paitients. It will reported as days.
drainage volume | 1 week
  This index will record the total volume from drainage tube after operation. It will reported as ml.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, Principal Investigator — Xi'an Jiaotong University Second Affiliated Hospital
Locations (1):
- Department of General Surgery , Second Afﬁliated Hospita l, Xi'an Jiaotong Universi ty School of Medicine, Xi'an, China

REFERENCES:
- [Derived] Liu Y, Wang J, Chen S, Lv H, Yu S, Ran X, Gao N, Sun Y, Cao G. Preliminary report on a novel technique for endoscopic transaxillary thyroidectomy: a case-control study. Int J Surg. 2024 Feb 1;110(2):654-659. doi: 10.1097/JS9.0000000000000885. PMID 37983762